CLINICAL TRIAL: NCT00273598
Title: Comparing the Moss Miami and Universal Spinal Instrumentation Systems for the Treatment of Adolescent Idiopathic Scoliosis
Brief Title: Comparing Two Instrumentation Systems for the Treatment of Adolescent Scoliosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Synthes Canada (Industry); DePuy-Acromed, Inc. (Industry); Johnson & Johnson (Industry)
Responsible Party: Principal Investigator, James Wright, Surgeon-in-Chief & Chief of Perioperative Services, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0019970040
Record Dates: First submitted 2006-01-04; First posted 2006-01-09 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Scoliosis
Keywords: Scoliosis; spinal disease; pediatrics; Adolescents; Universal Spinal Instrumentation System; Moss Miami Spinal Instrumentation System; Orthopedic Surgery
MeSH Terms: conditions — Scoliosis; Spinal Diseases

INTERVENTIONS:
Procedure: Moss Miami Spine Instrumentation System
Procedure: Universal Spine Instrumentation System

SUMMARY:
Idiopathic scoliosis affects 2-5% of adolescents. This study will compare the quality of life, functional outcome, cosmetic result, and the correction of spinal deformity of two instrumentation systems for the treatment of adolescent idiopathic scoliosis.

ELIGIBILITY:
Inclusion Criteria:

* Age 8-18 years
* Diagnosis of idiopathic scoliosis requiring posterior instrumentation and fusion(including those also requiring anterior release with or without anterior instrumentation) who could receive either the USS or the Moss Miami system
* Patients with scoliosis and an incidental finding of conus < L1-2 disc level, provided they have no symptoms or signs
* Patients with scoliosis and an incidental finding of a small syrinx (provided the syrinx is non-progressive and does not require neurosurgical treatment)
* Patients with non-progressive spondylolysis

Exclusion Criteria:

* Spinal cord abnormalities with any neurologic symptoms or signs
* Spinal cord lesions requiring neurosurgical interventions, such as hydromyelia requiring Arnold Chiari decompression
* Primary muscle diseases, such as muscular dystrophy
* Neurologic diseases (e.g. Charcot-Marie Tooth, Guillain-Barre syndrome, cerebral palsy, or spina bifida, etc.)
* Primary abnormalities of bones(e.g. osteogenesis imperfecta)
* Congenital scoliosis

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 126
Dates: Start 1997-09; Study Completion 2002-09 (Actual)

PRIMARY OUTCOMES:
- Quality of life at two years post-surgery, as measured by the self-report Quality of Life Profile for Spinal Disorders

SECONDARY OUTCOMES:
Physical function
Deformity, based on clinical exam and spinal radiographs
Clinicians' ratings of clinical photographs
Surgical outcomes, as measured by blood transfusions, duration of surgery,and length of hospitalization
Surgeons' global satisfaction with the instrumentation system
Complications of treatment (infection, loss of fixation, neurologic damage, and non-union)

CONTACTS AND LOCATIONS:
Overall Officials: James G Wright, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Background] Wright JG, Donaldson S, Howard A, Stephens D, Alman B, Hedden D. Are surgeons' preferences for instrumentation related to patient outcomes? A randomized clinical trial of two implants for idiopathic scoliosis. J Bone Joint Surg Am. 2007 Dec;89(12):2684-93. doi: 10.2106/JBJS.F.00720. PMID 18056501